CLINICAL TRIAL: NCT00139139
Title: A Blinded Randomized Comparative Study of Hepatitis A Vaccine and Immune Globulin for Postexposure Prophylaxis for Hepatitis A Disease
Brief Title: A Study to Compare the Efficacy of Hepatitis A Vaccine and Immune Globulin When Given After Exposure to Hepatitis A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Michigan (Other); Ministry of Health, Kazakhstan (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCID-2643; ASPHS196421/21
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis A
Keywords: hepatitis A; hepatitis A vaccine; immune globulin
MeSH Terms: conditions — Hepatitis A; Hepatitis | interventions — Hepatitis A Vaccines

INTERVENTIONS:
Biological: Hepatitis A vaccine

SUMMARY:
Immune globulin is effective about 85% of the time in preventing hepatitis A in people who have been exposed, if it is given within 14 days of exposure. Several lines of evidence suggest that hepatitis A vaccine might also be effective in this setting, and vaccine has the advantage of providing long term protection. In this study, we compare how well immune globulin and hepatitis A vaccine work in preventing clinical hepatitis A in household contacts of persons with the disease. The study's hypothesis is that the the proportion of exposed household contacts who receive hepatitis A vaccine within 14 days of exposure and develop hepatitis A disease will be similar to the proportion of exposure household contacts who receive immune globulin within 14 days of exposure and develop hepatitis A disease.

DETAILED DESCRIPTION:
Title: An Epidemiologic Study of Hepatitis A Vaccine for Postexposure Prophylaxis Clinical Phase: Investigation of an application unrelated to original approved use.

Primary Objective: To compare the clinical efficacy of vaccine and IG in the prevention of confirmed hepatitis A disease when given within 14 days of exposure to a confirmed case of hepatitis A disease.

Primary Hypothesis: The proportion of initially seronegative subjects who receive vaccine within 14 days of exposure to an index case of hepatitis A disease and who have onset of a confirmed case of hepatitis A disease within 56 days of exposure will be similar to the proportion of initially seronegative subjects who receive IG within 14 days of exposure to an index case and who have onset of a confirmed case of hepatitis A disease within 56 days of exposure. The date of exposure is defined as the date of onset of clinical symptoms in the index case.

(The statistical methods to examine this hypothesis require computing the relative risk, and corresponding 90% confidence interval, of confirmed hepatitis A disease among those receiving vaccine compared to those receiving IG, within 14 days of exposure. Inference of similarity involves examining the upper bound of this confidence interval and translating this RR bound into a lower bound of the 90% confidence interval for vaccine efficacy. Translation from relative risk to efficacy depends on an assumption of the point estimate of the efficacy of IG, based on historical data, the particular design of this study and assumptions regarding how transmission of hepatitis A virus occurred in the study population.) Study Design and Duration: Randomized, double-blinded, comparative, experimental epidemiologic study. Study will be conducted among exposed contacts 2-40 years of age in the household exposure group and is expected to last 18 months.

Sample Size: Enrollment will continue until 44 hepatitis A cases in randomized subjects are observed. Assuming a 30% secondary attack rate in evaluable, confirmed contacts of index cases and a 90% efficacy rate of IG, to observe 44 laboratory-confirmed cases of hepatitis A, 1468 randomized subjects will need to be evaluable (734/group). Evaluable is defined as seronegative at baseline and with clinical follow-up data at Day 56. Assuming 90% of subjects have follow-up data and 45% of subjects are seronegative at baseline, 4067 subjects ages 2 to 40 years must be randomized (2038/group). The actual enrollment may be different based on validity of these assumptions.

Dosage and Route: Within an exposed group, subjects will be randomized to receive either hepatitis A vaccine, VAQTA™, or immune globulin (IG) intramuscular (IM). Clinical material will be administered by unblinded study personnel but subjects will not be told which clinical material is being administered. The unblinded personnel will not be involved with any other study procedures for that exposed group. Syringes will be masked to avoid any possible chance at subject unblinding. The dose of VAQTA™ to be used will depend on the subject's age. Persons 2 to 18 years of age will receive a 25-U dose of VAQTA™ administered intramuscularly in the arm in a 0.5 mL volume. Persons 19 to 40 years of age and less than or equal to 75 kg in weight will receive a 50-U dose of VAQTA™ administered intramuscularly in the arm in a 1.0 mL volume. Persons 19 to 40 years of age and greater than 75 kg in weight will receive a 50-U dose of VAQTA™ (administered as two 25-U doses) administered intramuscularly with 0.5 mL in each arm. Persons 2 to 18 years of age will receive IG in one arm; persons 19 to 40 years of age and less than or equal to 75 kg in weight will receive IG in one arm; and persons 19 to 40 years of age and greater than 75 kg in weight will receive IG with the total dose equally divided between each arm. All persons randomized to receive IG will receive a dose of 0.02 mL/kg of body weight, up to a maximum of 1.5 mL for those less than or equal to 75 kg in weight and 3.0 mL for those greater than 75 kg in weight. All subjects less than or equal to 75 kg will receive 1 injection and only subjects 19 to 40 years of age and greater than 75 kg will receive 2 injections.

Efficacy Measurements: The primary measurement variable for efficacy is the proportion of subjects with confirmed hepatitis A disease (hepatitis A IgM positive or serum or stool PCR positive for HAV RNA and ALT twice the upper limit of normal with 1 or more of the clinical signs/symptoms of hepatitis A disease).

Safety Measurements: Subjects will be evaluated for serious or unusual reactions throughout the study period. The rate of serious adverse experiences in each group will be compared.

Data Analysis: In this study, efficacy comparisons will be made by estimation of the relative risk of laboratory-confirmed clinical hepatitis A in the vaccine group compared to the IG group. The relative risk is calculated as follows:

* where PV and PIG are the incidence rates of secondary cases of confirmed hepatitis A disease in the vaccine and immune globulin treatment groups, respectively.

The primary analysis will be performed at the one-sided ɑ=0.05 level and examine the upper bound of the 90% confidence for the relative risk of vaccine versus IG. A secondary efficacy analysis will adjust for the exposure group in the estimation of the relative risk.

The sample size and power are based upon a fixed number of events design assuming equal incidence rates in both the IG and vaccine populations and a one-sided significance level of ɑ=0.05, and were calculated under the following testing hypotheses: Ho: PV / PIG ≥3.0 versus Ha: PV / PIG <3.0. This is equivalent to testing that the upper bound of the 90% confidence interval on the observed relative risk is <3.0. For a fixed accrual of 44 evaluable secondary cases of confirmed hepatitis A, the study has 95% power to rule out a relative risk of 3.0 or greater. If the total number of cases observed in this study is 44 and if no more than 27 (i.e., 61.4%) of the cases are in the vaccine group, there will be significant evidence to reject the above null hypothesis. If the total number of cases is larger than 44, the maximum number of cases in the vaccine group that can be observed and still declare success will increase accordingly.

An internal pilot will be performed in a blinded fashion when ~25% of the 28 cases have occurred. This assessment will be done to check the assumptions pertaining to the incidence rate that was used to calculate the projected enrollment. A new sample size projection based upon the incidence rate (total across treatment groups) that had been observed thus far will be calculated for planning/budgetary concerns.

In addition, an interim analysis is proposed for the primary endpoint for potential early study termination if there is overwhelming evidence that vaccine is less efficacious than IG. The Independent Data Monitoring Committee (IDMC) will be responsible for making the recommendation on whether or not to continue the study based on the results of the interim analysis and relevant safety data. The interim analysis will be performed when 14 (~50%) of the 28 expected cases of laboratory-confirmed clinical hepatitis A have been observed. Using the same assumptions that were used for the original power calculation, the probability of meeting the success criteria at the end of the study conditioned on the number of cases that were observed in the vaccine group for the interim analysis will be calculated. If the probability is 20% or greater that vaccine will meet the assumed statistical criteria by the end of the study, then the study will definitely continue. In addition, if after 12 months from study start, very few cases have been observed, the IDMC will assess the need for study termination.

ELIGIBILITY:
Inclusion Criteria: Exposure to an index case of hepatitis A within 14 days of onset of illness; at least 2 years and no more than 40 years of age at time of study entry; susceptible to hepatitis A; give informed consent or have informed consent given by a responsible parent/guardian -

Exclusion Criteria: history of hepatitis A; prior receipt of hepatitis A vaccine; receipt of immune globulin within 180 days before study entry; evidence of liver disease; receipt of any live virus vaccine within 21 days prior to study entry; moderate or severe intercurrent illness or axillary temperature of 37.5 degrees or higher at time of study entry; various other medical conditions;

-

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1500
Dates: Start 2003-09; Study Completion 2005-05

PRIMARY OUTCOMES:
clincal hepatitis A disease

SECONDARY OUTCOMES:
1) subclinical hepatitis A
2) asymptomatic hepatitis A virus infection, with hepatitis A virus viremia

CONTACTS AND LOCATIONS:
Overall Officials: Beth P Bell, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Sanitary EpidemiologyAuthority, Almaty, Kazakhstan

REFERENCES:
- [Derived] Victor JC, Monto AS, Surdina TY, Suleimenova SZ, Vaughan G, Nainan OV, Favorov MO, Margolis HS, Bell BP. Hepatitis A vaccine versus immune globulin for postexposure prophylaxis. N Engl J Med. 2007 Oct 25;357(17):1685-94. doi: 10.1056/NEJMoa070546. Epub 2007 Oct 18. PMID 17947390